CLINICAL TRIAL: NCT04687046
Title: A Real-World Evidence Study of JUVÉDERM VOLUX® Injectable Gel for Chin Enhancement in Chinese Adults
Brief Title: A Study of JUVÉDERM VOLUX® Injectable Gel for Chin Enhancement in Chinese Adults Using Real-World Evidence
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 1868-705-008
Record Dates: First submitted 2020-12-02; First posted 2020-12-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chin Retrusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 JUVÉDERM VOLUX® with 3D Imaging: Treatment will be determined according to the physician's experience and Directions for Use. Cohort 1 will have follow-up on-site visits, including 3D imaging, at Months 1, 3, 6, and 12.
  Interventions: Device: JUVÉDERM VOLUX®
- Cohort 2 JUVÉDERM VOLUX®: Treatment will be determined according to the physician's experience and Directions for Use. Cohort 2 will have follow-up on-site visits at Months 1 and 3 and follow-up telephone calls at Months 6 and 12.
  Interventions: Device: JUVÉDERM VOLUX®

INTERVENTIONS:
Device: JUVÉDERM VOLUX® — JUVÉDERM VOLUX® injectable gel

SUMMARY:
This study will collect effectiveness and safety data on JUVÉDERM VOLUX® Injectable Gel for Chin Enhancement in Chinese Adults based on real world data.

DETAILED DESCRIPTION:
There will be 30 participants selected who undergo 3D imaging before and after JUVÉDERM VOLUX® treatment for digital analysis assessments. Up to 90 participants enrolled either prospectively prior to JUVÉDERM VOLUX® treatment or retrospectively after JUVÉDERM VOLUX® treatment.

ELIGIBILITY:
Inclusion Criteria:

-Participant has chin retrusion seeking chin enhancement who have received or plan to receive VOLUX chin treatment in Hainan Boao Super Hospital.

Exclusion Criteria:

* History of hypersensitivity to lidocaine,HA, or Streptococcal protein
* History of tendency to develop hypertrophic scarring
* Untreated epilepsy or porphyria
* Current cutaneous inflammatory or infectious processes (eg, acne, herpes) in the treatment area
* Prior chin or jaw surgery, including cartilage grafts or implantation of any biomaterials
* Permanent filler, semi-permanent filler, or fat injected in the treatment area
* Temporary filler, other than VOLUX, injected in the treatment area within 12 months before enrollment
* Females who self-report current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants receive VOLUX treatment at Hainan Boao Super Hospital, with screening and follow-up visits at Hainan Boao Super Hospital or another hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Glabella-Subnasale-Pogonion (G-Sn-Pog) Angle | Baseline, Month 3

SECONDARY OUTCOMES:
Percentage of Responders based on the Investigator's Assessment of Improvement in the Chin and Jaw Area using the 5-point Global Aesthetic Improvement Scale (GAIS) | Month 3
  The Evaluating Investigator will assess the aesthetic improvement of the hands using the GAIS 5- point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Percentage of Responders based on the Participant's Assessment of Improvement in the Chin and Jaw Area using the 5-point GAIS | Month 3
  Participant will assess the aesthetic improvement of the hands using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
The presence and severity of ISRs (Injection Site Response) at scheduled follow-up visits | Month 1, 3, 6, and 12
  The number of patients who experienced ISRs
The number of Adverse Events (AEs) from physician observation and inquiry at scheduled follow-up visits | Month 1, 3, 6, and 12
  The number of patients who experienced AEs

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (1):
- Hainan Boao Super Hospital /ID# 235968, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=1868-705-008&Latitude=&Longitude=&LocationName=#additional-resources-section